CLINICAL TRIAL: NCT01711996
Title: The Correlation Between Renal Injury and Biomarkers in Pediatric Ureteropelvic Junction Obstruction Patients
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty in purchasing reagents and receiving consent from the subject
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0421
Record Dates: First submitted 2012-10-17; First posted 2012-10-23 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Ureteropelvic Junction Obstruction
Keywords: hydronephrosis; biopsy; biomarker
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- UPJO: 0-3 year old hydronephrosis patients without ureter dilatation who undergo pyeloplasty
- Hydronephrosis: 0-3 year old hydronephrosis patients without ureter dilatation who does not meet the indication of pyeloplasty
- Normal: 0-3 year old children without hydronephrosis

SUMMARY:
Urinary Neutrophil gelatinase associated lipocalin (NGAL) has been recently reported to be related with the degree of hydronephrosis in pediatric ureteropelvic junction obstruction (UPJO) patients. We are trying to analyze whether it is related with the grade of renal injury in UPJO patients.

ELIGIBILITY:
Inclusion Criteria:

<Group 1>

1. 0-3 year old patients with SFU grade 2 or more hydronephrosis without ureteral dilatation
2. needs pyeloplasty due to differential renal function (DRF)<40%, decreased DRF by more than 5%, development of urinary tract infection, development of urinary stone, and development of pain related with UPJO <Group 2>

1. 0-3 year old patients with SFU grade 3 or 4 hydronephrosis without ureteral dilatation 2. doesn't meet the above criteria for the indication of pyeloplasty <Group 3>

1. 0-3 year old children without any abnormality of urinary tract

Exclusion Criteria:

<Group 1>

1. patients with contralateral disease affecting DRF
2. history of previous urinary tract surgery
3. follow up loss before diuretic renogram performed at 6-12 months from operation <Group 2, 3>

1. patients with contralateral disease affecting DRF 2. history of previous urinary tract surgery

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group 1: 20 patients with UPJO undergo pyeloplasty Group 2: 20 patients with hydronephrosis who does not meet the indication of pyeloplasty Group 3: 20 normal control
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The level of urinary NGAL and the degree of renal injury | 6 month after operation
  Analysis of correlation between the level of urinary NGAL and the degree of renal injury

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Urological Science Institute, Yonsei University, Colleage of Medicine, Seoul, South Korea